CLINICAL TRIAL: NCT00560131
Title: Evaluation of Autonomic Cardiac Function in Patients With Complex Regional Pain Syndrome
Brief Title: Evaluation of Autonomic Cardiac Function in Patients With CRPS
Status: Completed | Type: Observational
Sponsor: Danish Pain Research Center (Other)
Other Study IDs: Cardiac function in CRPS
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: CRPS (Complex Regional Pain Syndromes)
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the autonomic cardiac function in patients with complex regional pain syndrome

DETAILED DESCRIPTION:
Tilt table testing in patients with complex regional pain syndrome: Effects on heart rate variability and baroreceptor sensitivity.

Primary outcome parameter: Autonomic cardiac function

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 or older.
* Pain > 3 months.
* Diagnosed with CPRS acc. to diagnostic research criteria (Harder et al., 2005).
* Inclusion of healthy subjects: age-, gender-, and BMI-matched.

Exclusion Criteria:

* Other significant disease affecting the parameters measured, including cardiovascular disease.
* Treatment with anticholinergics, sympathomimetics and parasympathomimetics, and alpha- and beta-adrenergics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-06; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Autonomic cardiac function | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Troels S Jensen, MD, DMSc, Study Chair — Danish Pain Research Center, Aarhus University Hospital
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark